CLINICAL TRIAL: NCT07269340
Title: The Effect of Mandala Painting During Chemotherapy on Anxiety, Nausea, and Comfort Levels
Brief Title: Mandala Painting During Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Seda Pehlivan, Associate professor, Uludag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TPDD-2025-2369
Record Dates: First submitted 2025-11-24; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-05

CONDITIONS: Mandala Painting; Chemotherapy; Vomiting; Anxiety; Comfort; Nursing Care
MeSH Terms: conditions — Vomiting; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mandala Painting (Experimental): Patients receiving chemotherapy for the first time will have mandala painting done during their chemotherapy treatment.
  Interventions: Other: mandala painting
- Control Group (No Intervention): The patients in this group will not receive any intervention and will receive standard treatment and care during chemotherapy.

INTERVENTIONS:
Other: mandala painting — art therapy: mandala painting
  Arms: Mandala Painting

SUMMARY:
In addition to managing drug side effects that arise during cancer treatment, maintaining the patient's psychosocial well-being is also very important. Therefore, the aim of this project is to examine the effect of mandala painting during chemotherapy on anxiety, nausea, and comfort levels. This project aims to reduce the negative effects of chemotherapy, such as nausea, anxiety, and decreased comfort, by distracting the patient's attention through the non-invasive and non-pharmacological practice of mandala coloring in patients undergoing chemotherapy.

Mandala painting is a distraction and positive focus practice. A limited number of studies conducted on cancer patients have shown that it reduces distress and improves psychological well-being. However, no study in the literature has comprehensively addressed the symptoms experienced by patients during chemotherapy, such as anxiety, nausea, intense stress, and impaired comfort. The research will be conducted on patients undergoing chemotherapy for the first time, and patients in the experimental group will engage in mandala coloring for at least 30 minutes. Data obtained from assessments conducted before and after chemotherapy will be compared with control group data. This project will provide a more comprehensive assessment of the effect of mandala painting, a non-pharmacological intervention, on the negative symptoms of patients undergoing chemotherapy for the first time.

In addition to its scientific contribution, it is believed that effective symptom management can contribute to patients' well-being. Furthermore, if nausea can be controlled, the need for antiemetics during treatment can be reduced. This will also contribute to reducing unwanted drug effects and lowering costs.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old,
* Receiving chemotherapy for the first time

Exclusion Criteria:

* Have a lower education level than secondary school (The STAI is appropriate for those who have at least a sixth-grade reading level),
* Diagnosed with psychiatric and neurological diseases,
* Diagnosed with dementia,
* Received chemotherapy treatment more than once,
* Planned to receive radiotherapy treatment together with chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Anxiety level | baseline, 60-120 minute
  Baseline and post-intervention anxiety level assessed by trained research nurse using Spielberg's State-Trait Anxiety Inventory (STAI). The test scores between 20 and 80, with higher scores indicating more generalized and stronger anxiety.

SECONDARY OUTCOMES:
Nausea level | baseline, 60-120 minute
  Baseline and post-intervention nausea level assessed by trained research nurse using VAS (0 to 10; 0 means no nausea,10 means severe nausea).
Satisfaction level | 60-120 minute
  Post-intervention satisfaction level assessed by trained research nurse using VAS (0 to 10; 0 means not satisfied, 10 means very satisfied).
Comfort level | baseline, 60-120 minute
  Baseline and post-intervention comfort level assessed by trained research nurse using Distress Thermometer (0 to 10; 0 means no distress,10 means extreme distress).

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Uludağ University, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No